CLINICAL TRIAL: NCT07004517
Title: The Study on the Accuracy of Peri-implant Probing and Related Influencing Factors
Status: Recruiting | Type: Observational
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-51
Record Dates: First submitted 2025-05-13; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Peri-Implantitis; Diagnosis
MeSH Terms: conditions — Peri-Implantitis; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with dental implant restorations: Consecutive patients were selected who were treated at the Department of Oral Implantology, Stomatology Hospital, School of Medicine, Zhejiang University, Hangzhou, China,
  Interventions: Diagnostic Test: peri-implant probing before and after crown removal

INTERVENTIONS:
Diagnostic Test: peri-implant probing before and after crown removal — Before removal of the prosthetic reconstruction:
  * Measurement of PPD-1: The PPDs at 6 site were measured as the distance from the mucosal margin to the base of the peri-implant pocket.
  * Measurement of BOP-1：Bleeding sites after gentle probing within 15s were recorded as BOP scores. A positive score (1 point) was recorded if bleeding was observed during either of probing assessment by two researchers.
  After removal of the prosthetic reconstruction, PPD-2 and BOP-2 were recorded following the same protocol.

SUMMARY:
The aim of the diagnostic accuracy study was to compare the diagnostic accuracy of probing depth before (PPD-1) and following (PPD-2) the removal of prothesis in identifying the presence of peri-implantitis and assess the factors influencing peri-implant probing.

DETAILED DESCRIPTION:
This study aims to design a diagnostic accuracy study to compare the peri-implant probing depth and bleeding on probing before and after crown removal. It will explore the impact of prosthetic design on the accuracy of peri-implant probing and its diagnostic accuracy, and provide clinical recommendations on whether the prosthesis should be removed prior to peri-implant probing.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years.
2. The implant has completed osseointegration and has undergone final restoration for at least one month.
3. The final restoration needs to be removed or retrieved for various reasons.

Exclusion Criteria:

* Patients with serious systemic diseases, severe intraoral infections, severe mental disorders, pregnancy/lactation in women, or other conditions that make oral treatment operations unsuitable.
* History of crown removal or re-restoration within the past month prior to the visit.
* The prosthesis has fallen off or is severely damaged and has lost its original form before the visit.
* The prosthesis cannot be completely removed.
* Refusal to participate in this study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For this study, the calculation was estimated considering the peri-implantitis prevalence at implant level, thealternative the area under the receiver operating characteristic curve 0.90 , a 5% alpha error and 90% power. Thus, the minimum required sample size was 83 subjects.
Sampling Method: Probability Sample
Enrollment: 83 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
probing depth | On the day of enrollment
  The PPDs at 6 site were measured as the distance from the mucosal margin to the base of the peri-implant pocket.

SECONDARY OUTCOMES:
bleeding on probing | On the day of enrollment
  Bleeding sites after gentle probing within 15s were recorded as BOP scores. A positive score (1 point) was recorded if bleeding was observed during either of probing assessment by two researchers.
Emergency angel | The X-ray examination will be completed on the day of enrollment
  The emergence angle was calculated as the angle between the implant long axis and a line tangent to the restoration. The measurements were repeated twice, and the mean was calculated for each mesial and distal interproximal surface.
Emergency profile | The X-ray examination will be completed on the day of enrollment
  Emergence profile was categorized as either concave, straight or convex.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Stomatology Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China